CLINICAL TRIAL: NCT02488707
Title: Outcomes of Transanal Minimally Invasive TME Versus Laparoscopic Intersphincteric Resection Techniques for Rectal Cancer After Initial Neoadjuvant Chemo-radiotherapy: Double Blinded Study
Brief Title: Minimally Invasive Sphincter Sparing Total Mesorectal Excision for Ultra-low Rectal Cancer After Initial Chemo-radiotherapy (MISS-TRICR).
Acronym: MISS-TRICR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Osama Mohammad Ali ElDamshety, associate lecturer of surgical oncology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MISS-TRICR
Record Dates: First submitted 2015-06-27; First posted 2015-07-02 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Rectal Cancer
Keywords: low rectal cancer; minimally invasive colorectal surgery; trans-anal endoscopic microsurgery; TEM; intersphincteric resection; ISR; subtotal intersphincteric resection; total intersphincteric resection; trans-anal trans-abdominal resection; laparoscopic intersphincteric resection; anal sphincter preservation; total mesorectal excision; TME; TATA; laparoscopic total mesorectal excision; external sphincter preservation; Neoadjuvant chemo-radiotherapy for rectal cancer; fit patients for minimally invasive surgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LISR group (Active Comparator): Cases which undergo rectal resection with laparoscopic intersphincteric resection.
  Interventions: Procedure: laparoscopic intersphincteric resection (LISR group)
- TAMIS Group (Active Comparator): Cases with rectal cancer which undergo Transanal minimally invasive Total mesorectal excision.
  Interventions: Procedure: Transanal minimally invasive Total mesorectal excision (TAMIS group)

INTERVENTIONS:
Procedure: laparoscopic intersphincteric resection (LISR group) — the patient undergo laparoscopic mesorectal excision with high inferior mesenteric vein ligation combined with transanal distal resection of the rectum
  Other Names: Laparoscopic total mesorectum excision with coloaanal anastomosis.
  Arms: LISR group
Procedure: Transanal minimally invasive Total mesorectal excision (TAMIS group) — Transanal minimally invasive total mesorectal excision assisted with minilaparoscopy to ligate the inferior mesenteric vessels and splenic flexure mobilization.
  Arms: TAMIS Group

SUMMARY:
A prospective study is planned for management of low rectal cancer with the aim of sphincter preservation and improving the oncological outcome of the patients, through comparing of both approaches minimally invasive techniques including transanal total mesorectal excision and laparoscopic intersphincteric resection.

DETAILED DESCRIPTION:
Ideal surgery for rectal cancer should not only obtain adequate radial and circumferential margins, but also preserve normal sphincter function.In 1990, the results of a 'close shave' at anterior resection were reported, suggesting that a resection margin of 1 cm or less produced an oncological outcome similar to that of a resection margin greater than 1 cm.

Sphincter preservation presents several advantages; The lower risk of intraoperative rectal perforation and positive circumferential margin than APR, the lower risk of damaging the pelvic branches of the pelvic autonomic nerve and The preservation of the body image that may increase quality of life.

Recently, the clinical outcome of intersphincteric resection (ISR) as a laparoscopic approach (laparoscopic ISR) has been reported, but laparoscopic ISR for patients with bulky low rectal cancer remains challenging particularly for T3 tumors in patients with a narrow pelvis, because of the difficulty in understanding the accurate anatomy of the small pelvic cavity, in dissecting the TME or the tumor specific mesorectal excision (TSME) plane, and in transecting the lower rectum safely. Moreover, numerous studies have demonstrated that laparoscopic techniques have many advantages in colorectal surgery compared with open surgery.

Although Radical resection is the gold standard for the treatment of rectal cancer, TEM offers the advantage of combining a minimally invasive technique with evident benefits in terms of postoperative morbidity and recovery, long-term functional outcomes and subsequently improved quality of life. Transanal Endoscopic Microsurgery (TEM) developed at 1984 and eliminated most of local transanal excision limitations and triggered a significant improvement in the local excision procedures of rectal lesions. While TEM became the 'gold standard' for the treatment of large rectal adenomas and early rectal cancer, there are special concerns about the lack of adequate lymphadenectomy.

Preoperative chemoradiation therapy is widely used to treat locally advanced rectal cancer to increase resectability, and to enhance sphincter preservation, local control and possibly, survival rates. Surgery is performed six to eight weeks after radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with low rectal cancer below 5 cm from the anal verge
* Fit (Medically and surgically) for laparoscopy.

Exclusion Criteria:

* Patient with massive abdominal adhesions
* Unfit for laparoscopy
* Unwilling to share in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Percent of Intraoperative and postoperative morbidity within 30 days starting from the time of the operation | within 30 days
Hospital stay | up to 30 days
  Hospital stay starting from the day of admission till discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Osama eldamshety, PhD, Principal Investigator — Assistant Lecturer of surgical oncology; Sherif Kotb, PhD, MD, Study Chair — Professor of surgical oncology; Adel Fathi, PhD, MD, Principal Investigator — Lecturer of surgical oncology
Locations (1):
- Oncology centre Of Mansoura University (OCMU), Al Mansurah, Dakahlia Governorate, Egypt